CLINICAL TRIAL: NCT04401189
Title: The Role of Circadian Rhythms in Cancer-Related Symptoms: A Prospective Controlled Chrono-Bio-Behavioral Observation Study
Brief Title: The Role of Circadian Rhythms in Cancer-Related Symptoms
Acronym: CHRONO
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Ali Amidi, Assistant Professor, Aarhus University Hospital
Other Study IDs: 2016-051-000001- 1731
Record Dates: First submitted 2020-04-19; First posted 2020-05-26 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Fatigue; Cognitive Impairment; Sleep; Depression; Quality of Life; Stress, Psychological; Inflammation; Circadian Rhythm Disorders; Cancer-Related Syndrome
Keywords: Breast cancer; Circadian rhythms disruption; Cancer-related symptoms
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Cognitive Dysfunction; Depression; Stress, Psychological; Inflammation; Chronobiology Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples for melatonin. Blood samples for inflammatory cytokines.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients
- Healthy controls

SUMMARY:
Emerging evidence indicates that circadian rhythms may be disrupted following cancer and its treatment, and that circadian rhythm disruption may be an underlying pathophysiological mechanism of cancer- and cancer treatment-related symptoms (CRS) such as fatigue, sleep disturbance, cognitive impairment, and depressed mood. Given the detrimental effect of CRS on cancer survivors' quality of life, and a pressing demand for effective interventions to treat CRS, there is a need for a comprehensive examination of circadian disruption related to cancer and its treatment, and its association with CRS. The study will prospectively examine circadian rhythms and a CRS composite score in recently diagnosed breast cancer patients from prior to surgery or chemotherapy to 12 months later. A matched healthy control group will serve as a comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early breast cancer scheduled for surgery and chemotherapy (neoadjuvant or adjuvant) at Aarhus University Hospital (AUH).
* The healthy control group will consist of an age-matched sample of participants with no history of cancer.

Exclusion Criteria:

* Pregnancy
* Shift-work
* Melatonin supplementation
* Insufficient Danish proficiency
* Previous cancer diagnosis except for treated non-melanoma skin cancer
* Confounding diagnosed or suspected psychiatric or medical conditions that might significantly contribute to the CRS or symptoms/diagnoses resembling them (other than those caused by cancer or its treatment) such as seasonal affective disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients. Controls will be healthy volunteers of cancer-free women matched on age.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Cancer related symptoms composite score change | Change from baseline to time 2 (an average of 1 month)
  A composite score will be calculated based on measures of fatigue, sleep, cognition, and depression as described under secondary outcomes
Cancer related symptoms composite score change | Change from baseline to time 3 (an average of 6 months)
  A composite score will be calculated based on measures of fatigue, sleep, cognition, and depression as described under secondary outcomes
Cancer related symptoms composite score change | Change from baseline to time 4 (through study completion, an average of 1 year)
  A composite score will be calculated based on measures of fatigue, sleep, cognition, and depression as described under secondary outcomes
Circadian Activity Rhythms change | Change from baseline to time 2 (an average of 1 month)
  Rest/wake activity recorded with wrist actigraphy
Circadian Activity Rhythms change | Change from baseline to time 3 (an average of 6 months)
  Rest/wake activity recorded with wrist actigraphy
Circadian Activity Rhythms change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Rest/wake activity recorded with wrist actigraphy
Circadian skin temperature change | Change from baseline to time 2 (an average of 1 month)
  Distal skin temperature recorded with wrist actigraphy
Circadian skin temperature change | Change from baseline to time 3 (an average of 6 months)
  Distal skin temperature recorded with wrist actigraphy
Circadian skin temperature change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Distal skin temperature recorded with wrist actigraphy
Dim light melatonin onset change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Melatonin based on saliva samples

SECONDARY OUTCOMES:
Cognitive functioning change | Change from baseline to time 3 (an average of 6 months)
  Standard neuropsychological test battery
Cognitive functioning change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Standard neuropsychological test battery
Cancer-related fatigue change | Change from baseline to time 2 (an average of 1 month)
  FACIT fatigue
Cancer-related fatigue change | Change from baseline to time 3 (an average of 6 months)
  FACIT fatigue
Cancer-related fatigue change | Change from baseline to time 4 (through study completion, an average of 1 year)
  FACIT fatigue
Sleep change | Change from baseline to time 2 (an average of 1 month)
  Objective sleep recorded with wrist actigraphy
Sleep change | Change from baseline to time 3 (an average of 6 months)
  Objective sleep recorded with wrist actigraphy
Sleep change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Objective sleep recorded with wrist actigraphy
Inflammatory markers change | Change from baseline to time 3 (an average of 6 months)
  Proinflammatory cytokines known to mediate chronic inflammatory processes. Extracted from blood samples.
Inflammatory markers change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Proinflammatory cytokines known to mediate chronic inflammatory processes. Extracted from blood samples.
Stress change | Change from baseline to time 2 (an average of 1 month)
  Perceived Stress Scale (PSS)
Stress change | Change from baseline to time 3 (an average of 6 months)
  PSS
Stress change | Change from baseline to time 4 (through study completion, an average of 1 year)
  PSS
Sleep quality change | Change from baseline to time 2 (an average of 1 month)
  Pittsburgh sleep quality index
Sleep quality change | Change from baseline to time 3 (an average of 6 months)
  Pittsburgh sleep quality index
Sleep quality change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Pittsburgh sleep quality index
Insomnia change | Change from baseline to time 2 (an average of 1 month)
  Insomnia Severity Index
Insomnia change | Change from baseline to time 3 (an average of 6 months)
  Insomnia Severity Index
Insomnia change | Change from baseline to time 4 (through study completion, an average of 1 year)
  Insomnia Severity Index
Self-reported cognitive functioning change | Change from baseline to time 2 (an average of 1 month)
  Functional Assessment of Cancer Therapy - Cognitive function issues (FACT-Cog)
Self-reported cognitive functioning change | Change from baseline to time 3 (an average of 6 months)
  FACT-Cog
Self-reported cognitive functioning change | Change from baseline to time 4 (through study completion, an average of 1 year)
  FACT-Cog
Depression change | Change from baseline to time 2 (an average of 1 month)
  Center for Epidemiologic Studies Depression Scale (CESD)
Depression change | Change from baseline to time 3 (an average of 6 months)
  CESD
Depression change | Change from baseline to time 4 (through study completion, an average of 1 year)
  CESD
Self-reported quality of life change | Change from baseline to time 2 (an average of 1 month)
  Short Form 36 (SF36)
Self-reported quality of life change | Change from baseline to time 3 (an average of 6 months)
  SF36
Self-reported quality of life change | Change from baseline to time 4 (through study completion, an average of 1 year)
  SF36

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No